CLINICAL TRIAL: NCT04576351
Title: The Norwegian Study of Nervous System Manifestations and Sequelae After COVID-19
Acronym: NeuroCovid
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: University Hospital, Akershus (Other); Haukeland University Hospital (Other); Helse Stavanger HF (Other Government); St. Olavs Hospital (Other); University Hospital of North Norway (Other); Vestre Viken Hospital Trust (Other); Sykehuset Telemark (Other Government); Sykehuset Innlandet HF (Other); Ostfold Hospital Trust (Other); The Hospital of Vestfold (Other); Sorlandet Hospital HF (Other Government); Nordlandssykehuset HF (Other); Møre og Romsdal Hospital Trust (Other)
Responsible Party: Principal Investigator, Anne Hege Aamodt, Senior Consultant, MD, PhD, Oslo University Hospital
Other Study IDs: 152727
Record Dates: First submitted 2020-09-10; First posted 2020-10-06 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Covid19
Keywords: neurology
MeSH Terms: conditions — COVID-19 | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: Sub cohort 1:
  Participants in the WHO NOR Solidarity multicenter trial on the efficacy of different anti-viral drugs in SARS CoV-2 infected patients.
  Eligibility: consenting adults (age ≥18) hospitalized with definite COVID-19 included in the WHO COVID-19 Study. Participants invited to join the study will be those who are admitted to a collaborating hospital; no wider recruitment efforts are expected.
  Interventions: Other: Observation
- 2: Sub cohort 2:
  Patients with COVID-19 and neurological symptoms related to COVID-19 admitted to the Norwegian Departments of Neurology or other relevant Departments (both hospitalized and outpatient visits) and persons with neurological symptoms participating in other COVID-19 studies and not already participating in the WHO NOR Solidarity multicenter trial.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — The study is a multi-center Norwegian prospective observational clinical study of the occurence of neurological, neuropsychological and psychiatric manifestations and sequelae in patients with COVID-19 at 6- and 12-months follow-up.

SUMMARY:
Neurologic, neuropsychological and neuropsychiatric symptoms, signs and diagnoses are increasingly being reported in COVID-19 patients. However, the extent and implications of such "NeuroCOVID" involvement, as well as blood and MRI biomarkers for neurological and psychiatric COVID-19-affection and treatments, warrants further studies. The investigator will perform a national study with clinical and biomarker assessments of NeuroCOVID in approximately 150 Norwegian patients, recruited from ongoing COVID-studies in Norway as well as from neurological departments in Norway. The investigator will define the burden of neurological, psychological and psychiatric complications of COVID-19 disease and identify clinical characteristics and biomarkers for both short- and long-term neurological treatment and rehabilitation. Blood samples for biomarker analyses, brain MRI, clinical neurological, neurophysiological and neuropsychological assessments will be performed at 6 and 12 moths after acute disease,

DETAILED DESCRIPTION:
Corona virus (CoV) may have deleterious effects on the nervous system. As the number of individuals infected by the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) is increasing, more and more neurological, neuropsychological and neuropsychiatric symptoms are being reported in COVID-19 patients. Neurologists and psychiatrist, in turn, may increasingly find themselves involved in caring for patients with the novel virus.

Sars-CoV-2 usually enter the body via the enzyme angiotensin converting enzyme 2 (ACE2) in alveolar cells in the lungs. However, ACE2 is expressed in a number of other tissues and cells, such as mucous membranes of the eyes, nose and oral cavity, neurons, glia cells and endothelial cells, including those in the brain, making it a potential target of the virus.

There are several possible mechanisms for nervous system affection in COVID-19. Firstly, transneuronal transport of viruses through the olfactory nerve to the brain can induce direct injury. Sars-CoV-2 has been detected in cerebrospinal fluid in patients with encephalitis and meningitis. A second type of injury may result from an excessive immune response in the form of a "cytokine storm". Cytokines can cross the blood-brain barrier and are associated with acute necrotizing encephalopathy. A third mechanism of nervous tissue damage results from unintended host immune response effects after an acute infection. Examples of this type of indirect CNS injury are Guillain-Barré syndrome (GBS) and brain and spine demyelination. A fourth mechanism is an indirect viral injury that results from the effects of systemic illness, hypoxia and in some cases hypercoagulability, a prominent feature of severe COVID-19. Most cases of COVID-19-related neurologic complications appear to fall into this category. Severely ill patients in the intensive care unit may develop neurologic symptoms such as encephalopathy, critical illness myopathy, and neuropathy. This is common in both COVID-19 and in other diseases.

There have been several reports of nervous system manifestations in COVID-19. In a retrospective study from Wuhan China with 214 consecutive hospitalized patients, 1/3 had neurologic manifestations and nearly one half of those with severe infection. Common central nervous system (CNS) symptoms were dizziness, headache, and impaired consciousness or symptoms of acute cerebrovascular disease. The most common peripheral nervous system (PNS) symptoms included impaired taste, smell, or vision, and nerve pain. Skeletal muscular injury symptoms were also frequently reported. COVID-19 patients with CNS symptoms had lower lymphocyte levels and platelet counts and higher blood urea nitrogen levels compared to their counterparts without CNS symptoms. This may be indicative of immunosuppression in patients with COVID-19 and CNS symptoms or it may be manifestations coexisting in the same patient. Systematic brain imaging and measurements of neuron- or brain-specific biomarkers may increase the knowledge regarding nervous system manifestations in COVID-19 but were not performed in this study. Case report series with types of CNS or PNS manifestations, such as ischemic or hemorrhagic stroke, Guillain Barré syndrome, encephalitis, meningitis and toxic hemorrhagic necrotizing encephalopathy have been described. Furthermore, post infection surveillance will be necessary to identify possible post-COVID neurologic syndromes.

Moreover, COVID-19 is a significant psychological stressor, which may in addition to the neurological manifestations contribute to neuropsychiatric and neuropsychological sequela. Past respiratory viral pandemics have been associated with neuropsychiatric symptoms that may arise acutely or after variable periods of time. The long-term effect on neuropsychological functioning and the prevalence of neuropsychiatric symptoms due to COVID-19 are currently unknown. However, patients with COVID-19 are at risk of developing delirium that may cause long term cognitive impairment. Furthermore, Sars-CoV-2 proteins have been shown to interact with human proteins in multiple aging-related processes and CNS symptoms in patients with COVID-19 may put them at risk of neurocognitive complications. Given the global burden of COVID-19, long term neurocognitive complications are of importance to recognize.

Previously anxiety, depression and trauma related symptoms have been associated with CoV outbreaks. In survivors of SARS-CoV-1 active psychiatric illnesses were diagnosed in more than 40%, (PTSD (54%), depression (39%), somatoform pain disorders (36%), panic disorder (32%) and OCD (15%)) post-infection compared to pre-infection prevalence of less than 3%, and more than 27% had fatigue symptoms. Moreover, antibodies against CoV have been found in both psychoses and affective disorders. However, it is not known to which extent neuropsychological and psychiatric symptoms and disorders after COVID-19 are related to the psychological stressor or to CNS sequela after Covid-19 or to both.

Our hypotheses in this project are:

1. Nervous system manifestations and neurological sequelae are common after COVID 19.
2. Biomarkers in blood can be used to assess neurological manifestations and sequelae in COVID-19 patients at 6- and 12-months follow-up.
3. Severe COVID-19 infection predicts neurological manifestations and sequelae at 6- and 12-months follow-up.
4. Psychiatric disorders, especially anxiety and depressive disorders, but also psychotic and somatoform disorders are common after COVID-19, either due to CNS sequelae or manifestation or to perceived distress/strain.
5. Neuropsychological sequelae are common after COVID-19 either due to CNS sequelae or manifestation or to perceived distress/strain.
6. Biomarkers and imaging findings can be used to predict neuropsychiatric manifestations after Covid-19 at 6- and 12- months follow up.
7. Biomarkers in blood and imaging findings can be used to predict neuropsychological manifestations after Covid-19 at 6- and 12- months follow up.
8. Severe COVID-19 infection predicts neuropsychiatric and psychiatric disorders at 6- and 12-months follow-up.
9. Severe COVID-19 infection predicts neuropsychological sequelae at 6- and 12-months follow-up.

ELIGIBILITY:
Sub cohort 1:

Inclusion Criteria:

* Consenting adults (age ≥18 years) hospitalized with definite COVID-19 included in the WHO: The NOR Solidarity multicenter trial on the efficacy of different anti-viral drugs in SARS CoV-2 infected patients and willingness to participate in the NeuroCOVID study.

Exclusion Criteria:

* If still alive, no willingness and ability to participate in all follow-up examinations.

Sub cohort 2:

Inclusion Criteria:

* Consenting adults (age ≥18 years) with COVID-19 and new neurological, neuropsychological or neuropsychiatric symptoms and/or signs or participants from other COVID-19 studies than the NOR Solidary Study.

Exclusion Criteria:

* If still alive, no willingness and ability to participate in all follow-up examinations.

All participants in both sub cohorts will after the visit by neurologists be assessed by neuropsychologists and psychiatrist at 6- and 12-month follow-up if the following criteria are fulfilled:

1. Sufficient Norwegian or English speaking in order to fulfill the tests.
2. MoCA score > 18.
3. Hospital has C-L psychiatrist/neuropsychologists that participate in the study or collaborate with C-L psychiatrist/psychiatrist/clinical psychologists at nearby hospitals.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sub cohort 1: Participants in the WHO NOR Solidarity multi-center trial on the efficacy of different anti-viral drugs in SARS CoV-2 infected patients.
  Sub cohort 2: Patients with COVID-19 and new neurological, neuropsychological or neuropsychiatric symptoms and/or signs admitted to the Norwegian Departments of Neurology or other relevant Departments (both hospitalized and outpatient visits) or participants from other COVID-19 studies than the NOR Solidarity Study.
  Number of participants: Based on the number of included participants in the NOR Solidarity trial and the number of infected individuals we are planning to include 150 participants in the NeuroCOVID-19 study.
Sampling Method: Non-Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of peripheral and central nervous affection | 6 months
  Rate of neurological manifestations of COVID-19
Rate of peripheral and central nervous affection | 12 months
  Rate of neurological manifestations of COVID-19
Rate of psychiatric disorders at 6-months follow-up | 6 months
  Rate of psychiatric disorders as manifestations of COVID-19
Rate of psychiatric disorders at 12-months follow-up | 12 months
  Rate of psychiatric disorders as manifestations of COVID-19
Neuropsychological function at 6-months follow up | 6 months
  Neuropsychological function at 6-months follow up months after COVID-19. MoCA with score > 18 are eligible to further testing. Neuropsychological testing cover the most important domains of cognitive function enabling valid test data across different functional domains
Neuropsychological function at 12-months follow up and change in function from 6 to 12 months. | 12 months
  Neuropsychological function at 12-months follow up months after COVID-19. When MoCA > 18 at 6 months, MoCA is not done at 12 months. Neuropsychological testing cover the most important domains of cognitive function enabling valid test data across different functional domains.

SECONDARY OUTCOMES:
Rate of stroke at 6-months follow up | 6 months
  Rate of stroke
Rate of stroke at 12-months follow up | 12 months
  Rate of stroke
Rate of death at 6-months follow-up | 6 months
  Rate of death
Rate of death at 12-months follow-up | 12 months
  Rate of death
Rate of peripheral nervous affection assessed by clinical neurological examination and/or EMG/neurography at 6-months follow-up | 6 months
  Rate of peripheral nervous affection assessed by clinical neurological examination and/or EMG/neurography
Rate of peripheral nervous affection assessed by clinical neurological examination and/or EMG/neurography at 12-months follow-up | 12 months
  Rate of peripheral nervous affection assessed by clinical neurological examination and/or EMG/neurography
Rate of myopathy at 6-months follow-up | 6 months
  Rate of myopathy
Rate of myopathy at 12-months follow-up | 12 months
  Rate of myopathy
Rate of brain MRI pathology at 6-months follow-up | 6 months
  Rate of brain MRI pathology
Rate of brain MRI pathology at 12-months follow-up | 12 months
  Rate of brain MRI pathology
Levels of serum neurofilaments at 6-months follow-up | 6 months
  Levels of serum eurofilaments
Levels of serum neurofilaments at 12-months follow-up | 12 months
  Levels of serum neurofilaments
Rate of post-COVID neurological, cognitive or neuropsychiatric manifestations in the treatment arms at 6-months follow-up | 6 months
  Rate of post-COVID neurological, cognitive or neuropsychiatric manifestations in the treatment arms
Rate of post-COVID neurological, cognitive or neuropsychiatric manifestations in the treatment arms at 12-months follow-up | 12 months
  Rate of post-COVID neurological, cognitive or neuropsychiatric manifestations in the treatment arms
Duration of hospital and rehabilitation stay | 6 months
  Duration of hospital and rehabilitation stay at 6-months follow up
Duration of hospital and rehabilitation stay | 12 months
  Duration of hospital and rehabilitation stay at 12-months follow up

CONTACTS AND LOCATIONS:
Overall Officials: Anne Hege Aamodt, MD, PhD, Principal Investigator — Oslo University Hospital; Hanne F Harbo, MD,PhD,Prof, Study Director — Oslo University Hospital
Locations (15):
- Norway (15):
  - Sørlandet Hospital Trust, Arendal
  - Haukeland University Hospital, Bergen
  - Nordlandssykehuset, Bodø
  - Vestre Viken Hospital Trust Drammen, Drammen
  - Østfold Hospital Trust Kalnes, Grålum
  - Sørlandet Hospital Trust, Kristiansand, Kristiansand
  - Innlandet Hospital Trust, Lillehammer
  - Akershus University Hospital, Lørenskog
  - Møre og Romsdal Hospital Trust, Molde
  - Oslo University Hospital, Oslo
  - Ostfold Hospital Trust, Sarpsborg
  - Skien Hospital, Skien
  - Stavanger University Hospital, Stavanger
  - University Hospital of North Norway, Tromsø
  - St. Olav Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aamodt AH, Ueland T, Boldingh M, Bezgal BE, Argren MB, Dunne CA, Otterdal K, Gregersen I, Bjerkeli V, Michelsen AE, Husoy A, Morsund AH, Devik K, Poole AC, Gjendemsjo KB, Schluter K, Mathisen SM, Aalstad-Johansen M, Skattor TH, Sonnervik J, Boye TB, Popperud TH, Hogestol EA, Harbo HF, Lund-Johansen F, Aukrust P, Tronvik E, Dahl TB, Halvorsen BE. Altered amyloid plasma profile in patients with disabling headaches after SARS-CoV-2 infection and vaccination. BMJ Neurol Open. 2025 Aug 26;7(2):e001013. doi: 10.1136/bmjno-2024-001013. eCollection 2025. PMID 40881041